CLINICAL TRIAL: NCT06847334
Title: A Multicentre, Randomized, Double-Blind, Parallel-Controlled Integrated Phase I/III Clinical Study to Evaluate the Efficacy, Safety and Pharmacokinetic Profile of HLX17 Vs. Keytruda® (US-sourced Keytruda® and EU-sourced Keytruda®) in the First-Line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study to Compare the Efficacy, Safety, Immunogenicity, and Pharmacokinetic Profile of HLX17 Vs. Keytruda® in the First-Line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX17-NSCLC301
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
Keywords: Keytruda biosimilar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HLX17 group (Experimental): Recombinant anti-programmed death receptor-1- humanized antibody injection developed by Shanghai Henlius Biotech, Inc.
  Interventions: Drug: HLX17
- US-sourced Keytruda® group (Active Comparator): US-sourced Keytruda
  Interventions: Drug: US-sourced Keytruda®
- EU-sourced Keytruda® group (Active Comparator): EU-sourced Keytruda
  Interventions: Drug: EU-sourced Keytruda®

INTERVENTIONS:
Drug: HLX17 — HLX17 will be administered as IV infusion at a dose of 200mg on Day 1 of each 21-day cycle in combination with Carboplatin and Pemetrexed until loss of clinical benefit or up to 1 year.
  Arms: HLX17 group
Drug: US-sourced Keytruda® — US-sourced Keytruda® will be administered as IV infusion at a dose of 200mg on Day 1 of each 21-day cycle in combination with Carboplatin and Pemetrexed. After 24 weeks, all subjects in the US-Keytruda® group will receive HLX17 in combination with Pemetrexed until loss of clinical benefit or up to 1 year.
  Arms: US-sourced Keytruda® group
Drug: EU-sourced Keytruda® — EU-sourced Keytruda® will be administered as IV infusion at a dose of 200mg on Day 1 of each 21-day cycle in combination with Carboplatin and Pemetrexed until loss of clinical benefit or up to 1 year.
  Arms: EU-sourced Keytruda® group

SUMMARY:
This is a multicentre, randomized, double-blind, parallel-controlled integrated phase I/III clinical study to evaluate the similarity in efficacy, safety, PK profile, and immunogenicity of HLX17 vs. Keytruda®( US- and EU-sourced) in the first-line treatment of advanced non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This study includes three treatment groups. Patients will be randomly assigned at a 2:1:1 ratio to the HLX17, US-sourced Keytruda® and EU-sourced Keytruda® group to receive the treatment of IMPs in combination with Carboplatin Plus Pemetrexed until disease progression, initiation of new anti-tumor therapy, withdrawal of informed consent form, death, unacceptable toxicity, or up to 17 cycles (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV inoperable to surgery or radiotherapy (AJCC 8th edition) non-squamous NSCLC.
* Without any tumor activating EGFR mutation or ALK or ROS1 gene rearrangement.
* Have not received prior systemic treatment for their advanced/metastatic NSCLC.
* At least one measurable lesion as assessed by IRRC based on RECIST v1.1.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Have adequate organ function.

Exclusion Criteria:

* Subjects with NSCLC of other histopathological types, such as mixed adenosquamous carcinoma, and subjects with small cell lung cancer or neuroendocrine carcinoma.
* Subjects with other active malignancies within 5 years or at the same time prior to screening.
* Active central nervous system metastases.
* Known interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, and severe lung function abnormalities that may impede the investigators' diagnosis and management of drug-related pulmonary toxicity.
* Known active or suspected autoimmune diseases.
* History of immunodeficiency, including HIV antibody positive, active hepatitis B; or hepatitis C virus infections.
* Have received pembrolizumab or any other immune checkpoints inhibitors (PD-1, PD-L1, CTLA4, etc.) before screening.
* Pregnant or breastfeeding female.
* The investigator has a clear reason to believe that participation in this study would be detrimental to the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2025-04-27 (Estimated); Primary Completion 2027-04-09 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to 21 days (AUC0-21d) | Up to Day 21
Area under the serum concentration-time curve within a dosing interval at steady state (AUCss) | Up to 1 year
Best Objective Response Rate (BORR) assessed by Independent Radiology Review Committee (IRRC) based on RECIST v1.1 | up to week 24

SECONDARY OUTCOMES:
Maximum serum drug concentration (Cmax) after the first dose | Up to Day 21
Trough serum drug concentration (Ctrough) after the first dose | Up to Day 21
Area under the serum concentration-time curve from time 0 to infinity (AUC0-inf) after the first dose | Up to Day 21
Area under the serum concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCex) after the first dose | Up to Day 21
Time to reach maximum serum drug concentration (Tmax) after the first dose | Up to Day 21
Elimination half life (t1/2) after the first dose | Up to Day 21
Volume of distribution during terminal phase (Vz) after the first dose | Up to Day 21
Total clearance (CL) after the first dose | Up to Day 21
Mean residence time (MRT) after the first dose | Up to Day 21
Maximum serum drug concentration at steady-state (Cmax, ss) | Up to 1 year
Trough serum drug concentration at steady-state (Ctrough, ss) | Up to 1 year
Average serum drug concentration at steady-state (Cave, ss) | Up to 1 year
Time to reach maximum serum drug concentration at steady-state (Tmax, ss) | Up to 1 year
Elimination half life at steady-state (t1/2, ss) | Up to 1 year
Volume of distribution at steady-state (Vss) | Up to 1 year
Total clearance at steady-state (CLss) | Up to 1 year
Accumulation ratio of AUC (Rac(AUC)) | Up to 1 year
Accumulation ratio of Cmax (Rac(Cmax)) | Up to 1 year
Objective response rate (ORR) assessed by IRRC (based on RECIST v1.1) | Up to Week 24
Objective response rate (ORR) assessed by Investigator (based on RECIST v1.1) | Up to Week 48
Duration of response (DOR) assessed by the investigator (based on RECIST v1.1) | Up to Week 48
Time to response (TTR) assessed by the investigator (based on RECIST v1.1) | Up to Week 48
Progression free survival (PFS) assessed by the investigator (based on RECIST v1.1) | Up to Week 48
Progression free survival rate (PFSR) assessed by the investigator (based on RECIST v1.1) | Up to Week 48
Overall survival (OS) | Up to 1 year
Overall survival rate (OSR) | Up to 1 year
Adverse events (AEs) | Up to Month 15
Serious adverse events (SAEs) | Up to Month 15
Incidence of anti-drug antibodies (ADAs). | Up to 1 year
Incidence of neutralizing antibodies (NAbs). | Up to 1 year

IPD SHARING:
Plan to Share IPD: No